CLINICAL TRIAL: NCT05629338
Title: Evaluation for the Safety of FrontlineODP™ in a Multidose Randomized Cohort Study Compared With PF24
Brief Title: Ascending Dose Study of FrontlineODP™ Spray Dried Plasma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Velico Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: IDE 27346
Record Dates: First submitted 2022-10-28; First posted 2022-11-29 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Coagulopathy; Hemorrhage
Keywords: dried plasma; coagulation function; plasmapheresis
MeSH Terms: conditions — Hemostatic Disorders; Hemorrhage

STUDY DESIGN:
Intervention Model Description: This study in healthy volunteers (n=24) is designed to assess the safety of infusing ascending doses of reconstituted autologous FrontlineODP in 1, 2, and 4 fixed-dose units. Subjects in Cohort 1 (n = 6) will receive 1 unit of FrontlineODP (Arm 1), which is approximately 200 mL. Subjects in Cohort 2 (n = 6) will receive 2 FrontlineODP units (Arm 2) (total volume of approximately 400 mL). Cohort 3 is a crossover design where subjects (n = 12) will be randomly assigned to receive either 4 units of FrontlineODP followed 14 days later by 4 units of PF24 (Arm 3 - ODPxPF24), or 4 units of PF24 followed 14 days later by 4 units of FrontlineODP (Arm 4 - PF24xODP), where each infusion has a total volume of approximately 800 mL.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For Cohorts 1 and 2, blinding is not necessary because subjects will only receive a single infusion of FrontlineODP. Cohort 3 subjects will be randomly assigned to a treatment sequence and will remain blinded to the study product they receive at each visit. Study participants, the Principal Investigators, the Independent Medical Monitor, and the Data Monitoring Committee will be blinded to the randomization treatment assignments throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Cohort 1 (Experimental): Subjects are to have sufficient plasma withdrawn during a single plasmapheresis collection in the range of 625 - 800 mL, depending on subject's weight and hematocrit, to allow re-infusion with 1 unit (200 mL) of autologous FrontlineODP.
  Interventions: Combination Product: Autologous Spray Dried Plasma
- Cohort 2 (Experimental): Subjects are to have sufficient plasma withdrawn during a single plasmapheresis collection, in the range of 625 - 800 mL, depending on subject's weight and hematocrit, to allow re-infusion with 2 units (400 mL) of autologous FrontlineODP.
  Interventions: Combination Product: Autologous Spray Dried Plasma
- Cohort 3 Arm 3 (Active Comparator): Subject plasma is withdrawn during 4 plasmapheresis collections, in the range of 625 - 800 mL per collection, a total of approximately 2500 - 3200 mL, depending on subject's weight and hematocrit, to allow re-infusion with 4 units of autologous FrontlineODP and 4 units of autologous control PF24. Subjects will receive in total 8 units of plasma over the course of 2 infusion visits. Subjects randomized to Arm 3 will receive 4 units of FrontlineODP during the first infusion visit, and following a 14 day washout period, they would receive 4 units of PF24 during a second visit.
  Interventions: Combination Product: Autologous Spray Dried Plasma
- Cohort 3 Arm 4 (Active Comparator): Subject plasma is withdrawn during 4 plasmapheresis collections, in the range of 625 - 800 mL per collection, a total of approximately 2500 - 3200 mL, depending on subject's weight and hematocrit, to allow re-infusion with 4 units of autologous control PF24 and 4 units of autologous FrontlineODP. Subjects will receive in total 8 units of plasma over the course of 2 infusion visits. Subjects randomized to Arm 4 will receive 4 units of PF24 during the first infusion visit, and following a 14 day washout period, they would receive 4 units of FrontlineODP during the second visit.
  Interventions: Combination Product: Autologous Spray Dried Plasma

INTERVENTIONS:
Combination Product: Autologous Spray Dried Plasma — Evaluation of the Safety of Ascending Doses of Autologous Spray Dried Plasma in Healthy Volunteers
  Other Names: FrontlineODP Unit; Frontline On Demand Plasma Unit

SUMMARY:
This study in healthy volunteers is designed to assess the safety of infusing increasing doses of spray dried plasma (FrontlineODP).

DETAILED DESCRIPTION:
This study in healthy volunteers is designed to assess the safety of infusing increasing doses of spray dried plasma (FrontlineODP). Volunteers will have their plasma collected, spray dried, and then rehydrated for infusion. Volunteers will be infused with their own (autologous) rehydrated plasma. Cohort 1 will receive 1 FrontlineODP unit that is rehydrated to approximately 200 mL. Cohort 2 will receive 2 FrontlineODP units of approximately 400 mL. Cohort 3 volunteers will receive 2 separate infusions of 4 units of approximately 800 mL of either FrontlineODP (experimental) or frozen plasma (PF24). Order of receipt of plasma product will be randomized with 14 days between infusion.

ELIGIBILITY:
Inclusion Criteria:

* Males and nonpregnant/nonbreastfeeding females
* For females, a minimum weight of 140 pounds and maximum weight of 220 pounds; for males, a minimum weight of 140 pounds and a maximum weight of 250 pounds
* Subject is 18 to 65 years of age, inclusive
* Subject self-reports that he or she feels well and healthy
* Subject scores ≥35 on the Duke Activity Status Index
* Subject is able to donate a unit of plasma by plasmapheresis based on the AABB Donor History Questionnaire with modifications indicated: subjects with history of travel, which puts them at risk for Creutzfeldt-Jakob Disease or malaria, are eligible to participate
* Subject has completed a vaccination course for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), with the final vaccine injection administered at least 2 weeks before enrollment
* Subject has read the educational materials on donating blood and has had his or her questions answered
* Subject is able and willing to provide written informed consent
* Females of childbearing potential should either be surgically sterile (hysterectomy or tubal ligation) or should use a highly effective medically accepted contraceptive regimen. Highly effective methods of birth control are defined as those which result in a low failure rate (ie, less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices, sexual abstinence, condoms with spermicide, or vasectomized partner
* All females must have a negative urine or serum pregnancy test
* Subject understands the English language

Exclusion Criteria:

* Subject has known liver, kidney, cardiovascular, neurologic, gastrointestinal, blood, endocrine/metabolic, autoimmune, or pulmonary disease, or treated or untreated hypertension
* Subject has cancer of any kind, under treatment or resolved
* Subject has known or past coagulopathy conditions
* Subject has any conditions, uses medications, etc. on the AABB medical deferral list
* Subject has a history of asthma (defined as use of a prescribed daily asthma controller medication or required asthma medication in the past 2 weeks)
* Subject has a previous diagnosis of stroke, deep vein thrombosis (DVT), venous or arterial thrombosis, blood clots, or transient ischemic attack
* Subject has a family history of venous or arterial thrombosis before the age of 50 years in first degree relatives (ie, biological parents, full siblings, or children)
* Subject has a D-dimer test result ≥0.5 FEU/mL
* Subject has a recent (within 1 year of Screening) history of an abnormal electrocardiogram of clinical significance as determined by the site PI
* Subject has known HIV or AIDS-related illness or received a positive test result for HIV infection
* Subject has a positive test result for HBV, hepatitis C virus (HCV), or human T-cell lymphotropic virus
* Subject has a history of significant treated or untreated mental health issues
* Subject is currently taking an antibiotic or another medication for an infection
* Subject has received aspirin or other platelet-inhibiting agents within 14 days of study donation and infusion visits. Prior and concomitant medication information will be recorded beginning 30 days before enrollment through the final follow-up visit
* Subject is currently using any medications for anticoagulant therapy
* Subject has used clotting factor concentrates(s) (eg, FVIIa)
* Subject has received blood or blood products within the past 12 months
* Subject has had concurrent headache and fever in the past week
* Subject has systolic blood pressure (current) greater than 140 mm Hg
* Subject has diastolic blood pressure (current) greater than 90 mm Hg
* Subject has an oral temperature greater than 100°F
* Subject has known hematocrit ≤39% for male donors and ≤38% for female donors
* Subject has a positive DAT result
* Subject has received any investigational agent within 1 month before treatment infusion for this study
* Subject is participating in any phase of any other investigational studies while participating in this study
* Subject is unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's return for follow-up visits as scheduled
* Subject has other unspecified reasons that, in the opinion of the site PI, make the subject unsuitable for enrollment
* Subject is institutionalized because of legal or regulatory order
* Subject has a positive urine drug screen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Occurrence of Treatment-Emergent Adverse Events (TEAEs) | Start of plasma infusion through 28 day follow up (Day 29).
  Conclusions about safety will be based on the occurrence of TEAEs in Cohort 1 (1 unit of FrontlineODP, 200 mL) and Cohort 2 (2 units of FrontlineODP, 400 mL).
Occurrence of Treatment-Emergent Adverse Events (TEAEs) | Start of first plasma infusion through 28 day follow up of the second infusion (Day 43).
  Conclusions about safety will be based on the occurrence of TEAEs in Cohort 3 with infusions of 4 units (800 mL) of FrontlineODP compared to 4 units (800 mL) of PF24.

SECONDARY OUTCOMES:
Changes in PT | Start of first plasma infusion through 28-day follow up of second infusion (Day 43).
  changes between pre-infusion baseline and 4 hours post-infusion values after infusion of 4 units of FrontlineODP compared with infusion of the same dose of PF24.
Changes in INR | Start of first plasma infusion through 28-day follow up of second infusion (Day 43).
  changes between pre-infusion baseline and 4 hours post-infusion values after infusion of 4 units of FrontlineODP compared with infusion of the same dose of PF24.
Changes in aPTT | Start of first plasma infusion through 28-day follow up of second infusion (Day 43).
  changes between pre-infusion baseline and 4 hours post-infusion values after infusion of 4 units of FrontlineODP compared with infusion of the same dose of PF24.
Changes in Factor I | Start of first plasma infusion through 28-day follow up of second infusion (Day 43).
  changes between pre-infusion baseline and 4 hours post-infusion values after infusion of 4 units of FrontlineODP compared with infusion of the same dose of PF24.
Changes in Factor II | Start of first plasma infusion through 28-day follow up of second infusion (Day 43).
  changes between pre-infusion baseline and 4 hours post-infusion values after infusion of 4 units of FrontlineODP compared with infusion of the same dose of PF24.
Changes in Factor V | Start of first plasma infusion through 28-day follow up of second infusion (Day 43).
  changes between pre-infusion baseline and 4 hours post-infusion values after infusion of 4 units of FrontlineODP compared with infusion of the same dose of PF24.
Changes in Factor VII | Start of first plasma infusion through 28-day follow up of second infusion (Day 43).
  changes between pre-infusion baseline and 4 hours post-infusion values after infusion of 4 units of FrontlineODP compared with infusion of the same dose of PF24.
Changes in Factor VIII | Start of first plasma infusion through 28-day follow up of second infusion (Day 43).
  changes between pre-infusion baseline and 4 hours post-infusion values after infusion of 4 units of FrontlineODP compared with infusion of the same dose of PF24.
Changes in Factor IX | Start of first plasma infusion through 28-day follow up of second infusion (Day 43).
  changes between pre-infusion baseline and 4 hours post-infusion values after infusion of 4 units of FrontlineODP compared with infusion of the same dose of PF24.
Changes in Factor X | Start of first plasma infusion through 28-day follow up of second infusion (Day 43).
  changes between pre-infusion baseline and 4 hours post-infusion values after infusion of 4 units of FrontlineODP compared with infusion of the same dose of PF24.
Changes in Factor XI | Start of first plasma infusion through 28-day follow up of second infusion (Day 43).
  changes between pre-infusion baseline and 4 hours post-infusion values after infusion of 4 units of FrontlineODP compared with infusion of the same dose of PF24.
Changes in D-dimer | Start of first plasma infusion through 28-day follow up of second infusion (Day 43).
  changes between pre-infusion baseline and 4 hours post-infusion values after infusion of 4 units of FrontlineODP compared with infusion of the same dose of PF24.
Changes in von Willebrand Ristocetin Cofactor (vWF:RCo) activity | Start of first plasma infusion through 28-day follow up of second infusion (Day 43).
  changes between pre-infusion baseline and 4 hours post-infusion values after infusion of 4 units of FrontlineODP compared with infusion of the same dose of PF24.
Changes in von Willebrand (vWF) antigen | Start of first plasma infusion through 28-day follow up of second infusion (Day 43).
  changes between pre-infusion baseline and 4 hours post-infusion values after infusion of 4 units of FrontlineODP compared with infusion of the same dose of PF24.
Changes in protein S | Start of first plasma infusion through 28-day follow up of second infusion (Day 43).
  changes between pre-infusion baseline and 4 hours post-infusion values after infusion of 4 units of FrontlineODP compared with infusion of the same dose of PF24.
Changes in protein C | Start of first plasma infusion through 28-day follow up of second infusion (Day 43).
  changes between pre-infusion baseline and 4 hours post-infusion values after infusion of 4 units of FrontlineODP compared with infusion of the same dose of PF24.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Popovsky, MD, Study Director — Velico Medical
Locations (3):
- United States (3):
  - Hoxworth Blood Center, Cincinnati, Ohio
  - Versiti Blood Center of Wisconsin, Milwaukee, Wisconsin
  - Spaulding Clinical Research LLC, West Bend, Wisconsin

IPD SHARING:
Plan to Share IPD: No